CLINICAL TRIAL: NCT01626391
Title: A Double-Blind, Placebo-Controlled, Randomised, 4-Week Safety and Tolerability Study of TRx0237 in Subjects With Mild to Moderate Alzheimer's Disease on Pre-Existing Stable Acetylcholinesterase Inhibitor and/or Memantine Therapy
Brief Title: Safety Study of TRx0237 in Patients Already Taking Medications for Mild and Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated for administrative reasons only.
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRx-237-008
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-06

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's Disease; TRx0237; Safety Study; AD
MeSH Terms: conditions — Alzheimer Disease | interventions — hydromethylthionine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRx0237 (Experimental)
  Interventions: Drug: TRx0237
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRx0237 — TRx0237 tablets 250 mg/day (given as 125 mg bid) for 4 weeks
  Arms: TRx0237
Drug: Placebo — Placebo tablets will be administered twice daily (b.i.d.) for 4 weeks. The placebo tablets include 4 mg of TRx0237 as a urinary and faecal colourant to maintain blinding; hence, the placebo group will receive a total of 8 mg/day of TRx0237.
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to assess the safety and tolerability of TRx0237 when taken at the same time as acetylcholinesterase inhibitors (i.e., donepezil, galantamine, or rivastigmine) and / or memantine to treat patients with mild to moderate Alzheimer's Disease.

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of all cause dementia and probable Alzheimer's disease (AD)
* Mini-Mental State Examination (MMSE) score of 14-26 (inclusive)
* Cognitive impairment present for at least 6 months
* Age ≤90 years
* Modified Hachinski ischaemic score of ≤4
* Females, if of childbearing potential, must use adequate contraception and maintain this use throughout participation in the study
* Patient is able to read, understand, and provide written informed consent
* Has one or more identified caregivers who are able to verify daily compliance with study drug and provide information on safety and tolerability; the caregiver(s) must also give consent to participate
* Currently taking an taking an acetylcholinesterase inhibitor and/or memantine; the subject must have been taking such medication(s) for ≥3 months. The dosage regimen must have remained stable for ≥6 weeks and it must be planned to remain stable throughout participation in the study.
* Able to comply with the study procedures

Exclusion Criteria:

* Significant central nervous system disorder other than Alzheimer's disease
* Patients in whom baseline MRI is contraindicated such as metal implants in head (except dental), pacemaker, and cochlear implant
* Significant focal or intracranial pathology that would lead to a diagnosis other than probable Alzheimer's disease
* Clinical evidence or history of stroke, transient ischemic attack, significant head injury or other unexplained or recurrent loss of consciousness
* Epilepsy
* Major depressive disorder, schizophrenia or other psychotic disorders, bipolar disorder, substance (including alcohol) related disorders
* Resides in a hospital or continuous care facility
* History of swallowing difficulties
* Pregnant or breastfeeding
* History of significant hematological abnormality or current acute or chronic clinically significant abnormality
* Abnormal serum chemistry laboratory value at Screening deemed to be clinically relevant by the investigator
* Clinically significant cardiovascular disease or abnormal assessments
* Pre-existing or current signs or symptoms of respiratory failure
* Concurrent acute or chronic clinically significant immunologic, renal, hepatic, or endocrine disease (not adequately treated) and/or other unstable or major disease other than Alzheimer's disease
* Prior intolerance to methylthioninium-containing drug or any of the excipients
* Treatment currently or within 3 months before Baseline with any of the following medications (unless otherwise noted):

  * Tacrine
  * Anxiolytics and/or sedatives/hypnotics (exceptions: sedation for MRI or occasional short-acting benzodiazepines, chloral hydrate, or zolpidem as needed at bedtime)
  * Antipsychotics (clozapine, chlorpromazine, thioridazine, or ziprasidone)
  * Carbamazepine
  * Drugs associated with methaemoglobinaemia (e.g., dapsone, local anesthetics such as benzocaine used chronically, primaquine and related antimalarials, sulfonamides)
  * Warfarin (and other Coumadin derivates such as phenprocoumon)
* Current or prior participation in a clinical trial of a drug, biologic, or device in which the last dose was received within 28 days prior to Baseline

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-09; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dale, MD, Principal Investigator — MAC Clinical Research
Locations (12):
- Germany (4):
  - Achim
  - Berlin
  - Leipzig
  - München
- United Kingdom (8):
  - Birmingham
  - Bradford
  - Crowborough
  - Duston
  - Oxford
  - Saint Leonards-on-Sea
  - Sheffield
  - Staffordshire

RESULTS

PARTICIPANT FLOW:
Groups:
- TRx0237: One 125-mg TRx0237 tablet administered twice daily (250 mg/day TRx0237)
- Placebo: One placebo tablet containing 4-mg TRx0237 administered twice daily (8 mg/day TRx0237)
Period: Overall Study
Arm/Group | TRx0237 | Placebo
Started | 5 | 4
Completed | 3 | 4
Not Completed | 2 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | TRx0237 | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.2 (8.7) | 74.3 (3.3) | 74.2 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 4 | 9
Anti-dementia Therapy [Number; unit: participants]
  AChEI | 5 | 4 | 9
  Memantine | 0 | 0 | 0
  Both | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of TRx0237 When Coadministered With an Acetylcholinesterase Inhibitor (AChEI) and/or Memantine
Description: This was assessed by the number of participants who experienced adverse events within each treatment group (TRx0237 versus placebo) during 8 weeks of treatment.
Time Frame: 8 weeks
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | TRx0237 | Placebo
Number analyzed (Participants) | 5 | 4
participants | 4 | 4

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: At every visit, each subject was asked if he or she has experienced any adverse events and safety evaluations (including vital signs, clinical laboratory tests, pulse co-oximetry, 12-lead ECGs, physical and neurological evaluations, Columbia Suicide Severity Rating Scale and serotonin syndrome assessments) were performed throughout the study
Arm/Group | TRx0237 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 4/5 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRx0237 (N=5) | Placebo (N=4)
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urobilinogen urine increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Troponin I increased (Investigations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Intentional self-injury (Psychiatric disorders) | 1 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 1 | 0
Tooth repair (Surgical and medical procedures) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days